CLINICAL TRIAL: NCT03236597
Title: Assessing the Effects Of Treadmill On Light Physical Activity, Sitting Time, And Cardiovascular Risk
Brief Title: Assessing the Effects Of Treadmill On LPA, Sitting Time, and Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY000000866
Record Dates: First submitted 2017-07-27; First posted 2017-08-02 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Sedentary Lifestyle; Risk Factor, Cardiovascular
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A within-person, cross-over design will be used. Fifteen participants will take part in two conditions: 1) the treadmill desk: this intervention will ask participants to use a treadmill desk for a minimum of 30min per day for four weeks; and 2) the usual desk condition: participants will use their current workstation, as is, for four weeks. Participants will be randomly assigned to their initial intervention condition after baseline measures have been collected. In addition to the two condition months, there will be a one-week baseline period (to collected information on habitual activity level at work).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Desk (No Intervention): participants will work at their usual desk for four weeks.
- Treadmill desk (Experimental): Participants will be asked to use a treadmill desk for a minimum of 30 minutes per day for four weeks (Participants will sign up for a total of 30 minutes each day). Additional time may be spent on the treadmill, time permitting (two treadmills will be available to up to 10 people over the four week period).
  Interventions: Other: Treadmill desk

INTERVENTIONS:
Other: Treadmill desk — A standing height desk with a treadmill attached.
  Other Names: ActiveStation Treadmill desks
  Arms: Treadmill desk

SUMMARY:
The purpose of this study is to:

1. Evaluate the relative efficacy of a treadmill desk intervention on light physical activity and sitting behaviors at work over four weeks;
2. Evaluate the relative efficacy of a treadmill desk intervention on the cardiovascular risk profiles (blood pressure, body weight, body fat percentage) over a four-week period.

DETAILED DESCRIPTION:
American workers spend 70-80% of their time at work sitting at a desk, working on a computer, talking on a telephone, and sitting in meetings. Traditional approaches to increase MVPA in the workplace may not be sustainable as they require deliberate and dedicated time away from work, and may be perceived as harmful to productivity. Sedentary behavior interventions, in contrast, do not interfere with daily tasks and productivity and require small but cumulative changes in posture and LPA throughout the workday.

Sedentary behavior interventions in the worksite, including those conducted by our team, have shown promising effects. Studies that have used multi-level approaches targeting individual, social, and environmental factors have been most effective. The most robust environmental support has been the use of sit-stand workstations, providing distinct opportunities for workers to reduce sitting while maintaining productivity. However, treadmill desks may provide an even greater opportunity to both reduce sitting and increase LPA during the workday. Thus, a pilot study is required to test the efficacy of this approach to reduce sitting and increase LPA in the workplace.

ELIGIBILITY:
Inclusion Criteria:

* Not currently pregnant or planning to become pregnant during the 11 week study period.
* Able to read and write in English.
* No current use of a sit/stand or treadmill desk.
* Work that is done in a predominately stationary position.
* Working at UMN West Bank Office Building at least 30 hours per week.
* Not currently meeting physical activity guidelines.
* No balance issues (i.e. healthy vestibular system)
* No contraindications to standing or walking
* Weight stable for the past 12 months.
* Taking no more than 3 prescription drugs, with stable dosage, over the past 12 months
* Answer of no to all Physical Activity Readiness-Questionnaire (PAR-Q) questions

Exclusion Criteria:

* Currently pregnant or actively trying to become pregnant during the 14 week study period.
* Unable to read and write in English.
* Working less than 30 hours per week.
* Currently meeting physical activity guidelines.
* Non-sedentary job.
* Current use of treadmill desk
* Any reported balance problems
* Anyone with contraindications to standing or walking
* Weight fluctuations of more than +/- 10% of their body weight in the past year
* Individuals taking more than 4 prescription drugs and/or unstable dosage of medications over the past 12 months if taking 3 or less.
* Answer of yes to any PAR-Q questions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2019-12-08 (Actual)

PRIMARY OUTCOMES:
Time spent sitting | 7-days
  The change in time spent sitting as measured by the ActivPAL, from baseline to the final week of each intervention condition
Time spent standing | 7-days
  The change in time spent standing as measured by the ActivPAL, from baseline to the final week of each intervention condition
Time spent moving | 7-days
  The change in time spent moving as measured by the ActivPAL, from baseline to the final week of each intervention condition

SECONDARY OUTCOMES:
Cardiovascular risk: Blood pressure | 7-days
  The change in the cardiovascular risk, as measured via blood pressure from baseline to the final week of each condition.
Cardiovascular risk: Body weight | 7-days
  The change in the cardiovascular risk, as measured via body weight from baseline to the final week of each condition.
Cardiovascular risk: Percent body fat | 7-days
  The change in the cardiovascular risk, as measured via percent body fat from baseline to the final week of each condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota West Bank Office Building, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD for all primary and secondary outcome measures will be made available upon request.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will become available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the Principal Investigator. Requestors will be required to sign a data access agreement.